CLINICAL TRIAL: NCT06987903
Title: Impact of a Perioperative Physical Exercise and Respiratory Physiotherapy Program on the Patient Undergoing Bariatric Surgery
Acronym: CAPS-OB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Responsible Party: Principal Investigator, Marta López Otero, Principal Investigator, Fundacin Biomedica Galicia Sur
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CAPS-OB
Record Dates: First submitted 2024-12-17; First posted 2025-05-23 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Bariatric Surgery and Physical Activity; Obesity/Therapy; Bariatric Surgery Complications; Bariatric Patients
Keywords: Bariatric surgery; Obesity; Respiratory physiotherapy; Exercise programme
MeSH Terms: conditions — Motor Activity; Obesity | interventions — Lead

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): Specific pre- and post-operative physical exercise and respiratory physiotherapy programme.
  Interventions: Procedure: Pre- and post-operative physical exercise programme; Procedure: Pre- and post-operative respiratory physiotherapy
- Arm 2 (No Intervention): Usual pre- and post-operative procedure without a specific exercise programme.

INTERVENTIONS:
Procedure: Pre- and post-operative physical exercise programme — Pre- and post-operative physical exercise programme during 4 weeks before bariatric surgery and during 8 weeks after bariatric surgery for arm 1 participants.
  A program will be designed according to the needs and preferences of the individual and will include:
  Aerobic exercise: Activities that mobilize large muscle groups for prolonged periods of time.Walking, running at a slow or moderate pace (especially on a treadmill), cycling, cycloergometer, etc. In addition, due to the characteristics of the patients, the recommended exercises will be of low impact.
  Strength exercise: Exercises of large muscle groups with intensities adapted to patients using body weight or elastic bands of different resistances.
  Flexibility exercise: Stretching exercises will be included during the warm-up and cool-down of each exercise session of the program.
  Arms: Arm 1
Procedure: Pre- and post-operative respiratory physiotherapy — Pre- and post-operative respiratory physiotherapy during 4 weeks before bariatric surgery and during 8 weeks after bariatric surgery for arm 1 participants.
  Breathing exercises:
  Abdomino-diaphragmatic respiratory control exercises, costo-diaphragmatic respiratory control exercises, costo-diaphragmatic breathing control exercises, exercises with costal expansion and arm elevation and breathing exercises with pursed lips in different positions.
  Incentive spirometry:
  Incentive spirometry with the performance of slow, deep breaths in a volumetric incentive device.
  Arms: Arm 1

SUMMARY:
The goal of this clinical trial is to see the impact of a physical exercise programme and respiratory physiotherapy before and after bariatric surgery in obese patients. The main questions it aims to answer are:

Could it help to avoid decompensation of underlying diseases? Could it reduce the risks associated with the intervention and the number of adverse effects during the postoperative period? Could it reduce the number of patients and encourage early discharge? How does exercise affect epigenetics in obese patients undergoing bariatric surgery? Can we correlate epigenectic markers obtained from tissue obtained by invasive procedures such as fat or muscle to those obtained by non-invasive methods such as blood and saliva samples? How does exercise affect the hepatic tissue in obese patients undergoing bariatric surgery? And are the any predictive markers in pre-exercise samples that can correlate with the evolution of liver diseases such asl NALFD or NASH?

Researchers will compare one group of subjects performing the exercise programme and respiratory physiotherapy and anoher group performing the normal activities of routine clinical practice.

Participants, who are on the surgical waiting list for bariatric surgery, will be assigned to one of the two groups. Participants in group 2 will follow the normal procedure before and after surgery. Participants in group 1 will be asked to do a exercise programme and respiratory physiotherapy before and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing bariatric surgery at the General and Digestive Surgery Department of the Álvaro Cunqueiro Hospital in Vigo.
* Be over 18 and under 69 years old.
* Sign the informed consent to participate in the study.

Exclusion Criteria:

* Patient's refusal to enter the study.
* Inability to comprehend participation in a study.
* Urgent interventions.
* Patients undergoing combined surgery with another surgical service.
* Patients who cannot read and write or are dependent on a legal representative.
* Patients on treatment for diabetes with GLP-1 agonists (glucagon-like peptide type 1 agonists) and/or SGLT2 inhibitors (sodium-glucose cotransporter type 2 inhibitors) whose dose is not stable in the last 3 months.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2026-05-07 (Estimated); Study Completion 2026-09-07 (Estimated)

PRIMARY OUTCOMES:
Total weight loss | From enrollment to the end of intervention at 8 weeks
  [(Preoperative weight - Weight at 8 weeks post-operative) / Preoperative weight]*100
Waist circumference | From enrollment to the end of intervention at 8 weeks
  Waist circumference measured in cm
Sex (at birth) | Once at the inclusion

SECONDARY OUTCOMES:
Comorbidities | 4 weeks before bariatric surgery
  It will indicate which comorbidities the patient has from a list with the following options:
  Hypertension, type 2 diabetes mellitus, dyslipidaemia, COPD, OSAS / OSHS, cardiovascular, GERD, arthropathy, infertility, neoplasias, psoriasis, hepatics, deppresion.
Age | 4 weeks before bariatric surgery
  Age in years
Concomitant medication | 4 weeks before bariatric surgery
  It will indicate which concomitant medication the patient has from a list with the following options:
  Anticoagulant, antiaggregant, stable GLP1 agonist.
Active smoking | 4 weeks before bariatric surgery
  Yes/No
Alcohol consumption | 4 weeks before bariatric surgery
  Alcohol consumption in UBEs or Units of alcohol
Previous abdominal surgeries | 4 weeks before bariatric surgery
  Yes/No
Previous bariatric interventions | 4 weeks before bariatric surgery
  Yes/No
Weight at inclusion | 4 weeks before bariatric surgery
  Kilograms
Height at inclusion | 4 weeks before bariatric surgery
  Metres
Impedanciometry | 4 weeks before bariatric surgery
  Fat mass, bone mass, muscle mass, intracellular and extracellular water mass.
ASA Score | 4 weeks before bariatric surgery
Baseline O2 Saturation | 4 weeks before bariatric surgery
  %
Blood glucose | From enrollment to the end of intervention at 8 weeks
  mg/dL
Haemoglobin A1c | From enrollment to the end of intervention at 8 weeks
  % Myokines and exerkines, lactate, insulin. Oxidative stress markers. DNA methylation profile and gene expression. Lipidomic and metabolomic profile.
Total protein | From enrollment to the end of intervention at 8 weeks
  g/dL Myokines and exerkines, lactate, insulin. Oxidative stress markers. DNA methylation profile and gene expression. Lipidomic and metabolomic profile.
Albumin | From enrollment to the end of intervention at 8 weeks
  g/dL Myokines and exerkines, lactate, insulin. Oxidative stress markers. DNA methylation profile and gene expression. Lipidomic and metabolomic profile.
Pre-Albumin | From enrollment to the end of intervention at 8 weeks
  mg/dL Myokines and exerkines, lactate, insulin. Oxidative stress markers. DNA methylation profile and gene expression. Lipidomic and metabolomic profile.
Cholesterol | From enrollment to the end of intervention at 8 weeks
  mg/dL Myokines and exerkines, lactate, insulin. Oxidative stress markers. DNA methylation profile and gene expression. Lipidomic and metabolomic profile.
Triglycerides | From enrollment to the end of intervention at 8 weeks
  mg/dL Myokines and exerkines, lactate, insulin. Oxidative stress markers. DNA methylation profile and gene expression. Lipidomic and metabolomic profile.
HDL Cholesterol | From enrollment to the end of intervention at 8 weeks
  mg/dL Myokines and exerkines, lactate, insulin. Oxidative stress markers. DNA methylation profile and gene expression. Lipidomic and metabolomic profile.
LDL Cholesterol | From enrollment to the end of intervention at 8 weeks
  mg/dL
AST (GOT) | From enrollment to the end of intervention at 8 weeks
  UI/L Myokines and exerkines, lactate, insulin. Oxidative stress markers. DNA methylation profile and gene expression. Lipidomic and metabolomic profile.
ALT (GPT) | From enrollment to the end of intervention at 8 weeks
  UI/L Myokines and exerkines, lactate, insulin. Oxidative stress markers. DNA methylation profile and gene expression. Lipidomic and metabolomic profile.
GGT | From enrollment to the end of intervention at 8 weeks
  UI/L Myokines and exerkines, lactate, insulin. Oxidative stress markers. DNA methylation profile and gene expression. Lipidomic and metabolomic profile.
Alkaline phosphatase | From enrollment to the end of intervention at 8 weeks
  UI/L Myokines and exerkines, lactate, insulin. Oxidative stress markers. DNA methylation profile and gene expression. Lipidomic and metabolomic profile.
LDH | From enrollment to the end of intervention at 8 weeks
  UI/L Myokines and exerkines, lactate, insulin. Oxidative stress markers. DNA methylation profile and gene expression. Lipidomic and metabolomic profile.
Iron | From enrollment to the end of intervention at 8 weeks
  µg/dL Myokines and exerkines, lactate, insulin. Oxidative stress markers. DNA methylation profile and gene expression. Lipidomic and metabolomic profile.
Transferrin | From enrollment to the end of intervention at 8 weeks
  µg/dL Myokines and exerkines, lactate, insulin. Oxidative stress markers. DNA methylation profile and gene expression. Lipidomic and metabolomic profile.
Transferrin saturation rate | From enrollment to the end of intervention at 8 weeks
  % Myokines and exerkines, lactate, insulin. Oxidative stress markers. DNA methylation profile and gene expression. Lipidomic and metabolomic profile.
Ferritin | From enrollment to the end of intervention at 8 weeks
  ng/mL
Vitamin B12 | From enrollment to the end of intervention at 8 weeks
  pg/mL Myokines and exerkines, lactate, insulin. Oxidative stress markers. DNA methylation profile and gene expression. Lipidomic and metabolomic profile.
Folic acid | From enrollment to the end of intervention at 8 weeks
  ng/mL
Lactate | From enrollment to the end of intervention at 8 weeks
  mmol/L Myokines and exerkines, lactate, insulin. Oxidative stress markers. DNA methylation profile and gene expression. Lipidomic and metabolomic profile.
Exerkines | From enrollment to the end of intervention at 8 weeks
  ng/mL Myokines and exerkines, lactate, insulin. Oxidative stress markers. DNA methylation profile and gene expression. Lipidomic and metabolomic profile.
Myokines | From enrollment to the end of intervention at 8 weeks
  ng/mL
IL | From enrollment to the end of intervention at 8 weeks
  pg/mL
Grip strength dynamometry | From enrollment to the end of intervention at 8 weeks
Goniometry | 4 weeks before bariatric surgery
  Joint goniometry of the main joints of the extremities (shoulder, elbow, wrist, hip, knee, ankle) will be performed to rule out important joint limitations that also require some type of adaptation in the exercise program.
Sit to stand Test | From enrollment to the end of intervention at 8 weeks
  5 repetitions
6' walk test | From enrollment to the end of intervention at 8 weeks
  Distance walked and Vo2max estimation
Walking speed test | From enrollment to the end of intervention at 8 weeks
  Time to cover 4 metres at usual pace.
IPAQ | From enrollment to the end of intervention at 8 weeks
  International Physical Activity Questionnaire. High, moderate, low.
ARISCAT | 4 weeks before bariatric surgery
  Score for Postoperative Pulmonary Complications. From 0 (Low risk) to 123 points (High risk)
Oral tolerance | Immediate postoperative period up to 12 hours after surgery
  (YES/NO)
Beginning of standing | Immediate postoperative period up to 12 hours after surgery
  (YES/NO)
Urinary catheterisation | Immediate postoperative period up to 12 hours after surgery
  (YES/NO)
Use of respiratory incentive | The first day after surgery
  (YES/NO)
EVA of level of subjetive pain felt | The first, second and third day after surgery
  Visual analog scale from zero (0) to ten (10). Zero being no pain at all, ten being the worst pain imaginable
Morbidity/complications | The fourth day after surgery
  (YES/NO)
Days from post-operative period to discharge | The fourth day after surgery
  Days
Emergency attendance in the first 30 days from discharge | 8 weeks after discharge
  (YES/NO)
Re-admission in General and Digestive Surgery Department | 8 weeks after discharge
  (YES/NO)
Re-intervention during re-admission | 8 weeks after discharge
  (YES/NO)
Average daily steps | 8 weeks after discharge
Adverse events during exercise | From enrollment to the end of intervention at 8 weeks
  Dizziness, pain, dyspnoea
Compliance with exercise programme. | 8 weeks after discharge
  Only in arm 1 participants. (0%, <50%, >50 - <100%, 100%)
EuroQol 5D (Quality of Life Questionnaire) | From enrollment to the end of intervention at 8 weeks
  Quality of Life Questionnaire. From 0 to 100, where 100 is the best possible health state.
Suter oral tolerance test | 8 weeks after discharge
  Questionnaire for assessment of food tolerance after bariatric surgery. From 1 to 27, where 27 is the best food tolerance.
Surgical Variable: Kind of approach | In bariatric surgery
  It will indicate which kind of approach from a list with the following options:
  Simple laparoscopy, 3D Laparoscopy, Single port, Reduced ports, Assisted robotics (DaVinci Xi), Laparotomy
Surgical Variable: number of trocars | In bariatric surgery
  Number of trocars
Surgical Variable: surgical technique | In bariatric surgery
  It will indicate which surgical technique from a list with the following options:
  Gastric bypass, Vertical gastrectomy, Nissen-Sleeve, SADI, Other
Surgical Variable: associated surgery | In bariatric surgery
  (YES/NO)
Surgical Variable: revision surgery | In bariatric surgery
  (YES/NO)
Surgical Variable: opioid-free anesthetic protocol (OFA) | In bariatric surgery
  (YES/NO)
Surgical Variable: Intraoperative pneumatic compression stockings | In bariatric surgery
  (YES/NO)
Surgical Variable: urinary catheterisation | In bariatric surgery
  (YES/NO)
Surgical Variable: intra-abdominal drainage | In bariatric surgery
  (YES/NO)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Alvaro Cunqueiro, Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No